CLINICAL TRIAL: NCT04409509
Title: A Phase 2, Multicenter, Double Blind, Randomized, Placebo-Controlled Study to Evaluate CSL312 in Coronavirus Disease 2019 (COVID 19)
Brief Title: Treatment With CSL312 in Adults With Coronavirus Disease 2019 (COVID-19)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSL312_COVID-19
Record Dates: First submitted 2020-05-28; First posted 2020-06-01 (Actual); Results first posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Coronavirus Disease 2019 (COVID-19)
Keywords: Prevention of respiratory failure
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CSL312 (Experimental): Garadacimab, Factor XIIa Antagonist Monoclonal Antibody administered intravenously
  Interventions: Biological: Garadacimab, Factor XIIa Antagonist Monoclonal Antibody
- Placebo (Placebo Comparator): CSL312 diluent administered intravenously
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Garadacimab, Factor XIIa Antagonist Monoclonal Antibody — Garadacimab, Factor XIIa Antagonist Monoclonal Antibody administered intravenously
  Arms: CSL312
Drug: Placebo — CSL312 diluent administered intravenously
  Arms: Placebo

SUMMARY:
This is a prospective, phase 2, multicenter, randomized, double blind, placebo controlled, parallel group study to assess the safety and efficacy of CSL312 administered intravenously, in combination with standard of care (SOC) treatment, in patients with Coronavirus disease 2019 (COVID 19)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Positive for severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) infection as determined using a molecular diagnostic test (reverse transcription polymerase chain reaction [RT-PCR] or equivalent) approved by regulatory authorities (including Food and Drug Administration or Brazilian Health Regulatory Agency) or allowed under an emergency use authorization within 14 days before Screening. If a false negative result is suspected, the SARS-CoV-2 test may be repeated within the Screening Period.
* Chest CT scan or X ray results confirming interstitial pneumonia
* Severe COVID 19 disease as evidenced by ≥ 1 of the following criteria at Screening including within 24 hours before Screening:

  * Respiratory frequency > 30 breaths per minute
  * SpO2 ≤ 93% on room air
  * Ratio of partial pressure of arterial oxygen to fraction of inspired oxygen (PaO2/FiO2) < 300
  * Ratio of Arterial oxygen saturation to fraction of inspired oxygen (SaO2/FiO2 ratio) < 218 (if PaO2/FiO2 ratio is not available)
  * Radiographic lung infiltrates > 50%

Exclusion Criteria:

* Currently enrolled, planning to enroll, or participated, within the last 30 days, in a clinical study requiring administration of an IP, including expanded access or compassionate use with the only exception being administration of convalescent plasma. Administration of IP is permitted only if an emergency use authorization has been granted (eg, remdesivir). Additionally, off label use of approved drugs (eg, anti IL 6/anti IL 6R) is also permitted.
* Pregnant or breastfeeding (female subjects)
* Intubated and require mechanical ventilation (including ECMO) at the time of randomization
* In the opinion of the investigator, the subject is expected to be intubated in the first 24 hours after IMP administration
* Has a Do-Not-Intubate (DNI) or Do-Not-Resuscitate (DNR) order
* In the opinion of the investigator, not expected to survive for > 48 hours after admission
* Presence of any of the following comorbid conditions prior to randomization and prior to SARS CoV 2 infection:

  * Severe heart failure (New York Heart Association Class IV)
  * End stage renal disease (Stage ≥ 4) or need for renal replacement therapy
  * Biopsy confirmed cirrhosis, portal hypertension, or hepatic encephalopathy
  * Malignancy (Stage IV)
  * Chronic lung disease requiring the use of oxygen at home
  * Active tuberculosis disease
* Active bleeding or a current clinically significant coagulopathy (eg, international normalized ratio [INR] > 1.5) or clinically significant risk for bleeding (eg, recent intracranial hemorrhage or bleeding peptic ulcer within the last 4 weeks)
* History of venous thrombosis, myocardial infarction or cerebrovascular event within 3 months, or a prothrombotic disorder (eg, antithrombin III, protein C or protein S deficiency)
* Known or suspected Grade 3 or 4 infusion-related reaction or hypersensitivity (per Common Terminology Criteria for Adverse Events [CTCAE]) to monoclonal antibody therapy, or hypersensitivity to the IMP or any excipients of the IMP
* Currently receiving a therapy not permitted during the study.
* Female subject of childbearing potential or fertile male subject either not using or not willing to use an acceptable method of contraception to avoid pregnancy during the study and for 90 days after receipt of the last dose of IMP
* Any clinical or laboratory abnormality or other underlying conditions (eg, psychological disorders, substance abuse) that would render the subject unsuitable for participation in the study, in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (14):
- United States (14):
  - Nova Clinical Research, LLC, Bradenton, Florida
  - Theia Clinical Research, LLC, St. Petersburg, Florida
  - MercyOne North Iowa Medical Center, Mason City, Iowa
  - Northeast Iowa Medical Education Foundation, Waterloo, Iowa
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Holy Name Hospital, Teaneck, New Jersey
  - Inspira Health Center Vineland, Vineland, New Jersey
  - Sisters of Charity Hospital/ St. Joseph's Campus, Buffalo, New York
  - Carolina Institute for Clinical Research, Fayetteville, North Carolina
  - Monument Health Clinical Research, Rapid City, South Dakota
  - PharmaTex Research, Amarillo, Texas
  - UT Health Science Center, McGovern Medical School, Houston, Texas
  - Inova Alexandria Hospital, Alexandria, Virginia

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider requests to share Individual Patient Data (IPD) from systematic review groups or bona-fide researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.
Supporting Information: Study Protocol, SAP
Time Frame: IPD requests may be submitted to CSL no earlier than 12 months after publication of the results of this study via an article made available on a public website.
Access Criteria: Requests may only be made by systematic review groups or bona-fide researchers whose proposed use of the IPD is non-commercial in nature and has been approved by an internal review committee.
  An IPD request will not be considered by CSL unless the proposed research question seeks to answer a significant and unknown medical science or patient care question as determined by CSL's internal review committee.
  The requesting party must execute an appropriate data sharing agreement before IPD will be made available.

REFERENCES:
- [Derived] Papi A, Stapleton RD, Shore PM, Bica MA, Chen Y, Larbig M, Welte T. Efficacy and Safety of Garadacimab in Combination with Standard of Care Treatment in Patients with Severe COVID-19. Lung. 2023 Apr;201(2):159-170. doi: 10.1007/s00408-023-00615-9. Epub 2023 Mar 31. PMID 37000214

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | CSL312
Started | 61 | 63
Completed | 48 | 43
Not Completed | 13 | 20
Not completed — Failure to meet randomization requirement | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Death | 11 | 10
Not completed — Non-compliance with study drug | 0 | 1
Not completed — Lost to Follow-up | 0 | 3
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Randomized by mistake | 0 | 1
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | CSL312 | Total
Number analyzed (Participants) | 61 | 63 | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 32 | 65
  >=65 years | 28 | 31 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (12.74) | 62.7 (14.61) | 62.5 (13.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 30 | 50
  Male | 41 | 33 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 14 | 24
  Not Hispanic or Latino | 48 | 48 | 96
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 7 | 13
  White | 49 | 44 | 93
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 3 | 9 | 12
Region of Enrollment [Number; unit: participants]
  United States | 61 | 63 | 124

OUTCOME MEASURES:

1. Primary Outcome: The Percent of Participants With Tracheal Intubation or Death Prior to Tracheal Intubation
Time Frame: From randomization to Day 28
Population: Intent-to-treat Analysis Set (ITT) comprises all subjects who were randomly assigned to treatment and who were assigned randomization numbers.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CSL312
Number analyzed (Participants) | 61 | 63
percentage of participants | 26.2 | 22.2

2. Secondary Outcome: Percent of Participants With Death From All Causes
Time Frame: From randomization to Day 28
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CSL312
Number analyzed (Participants) | 61 | 63
percentage of participants | 18.0 | 17.5

3. Secondary Outcome: Percent of Participants With Tracheal Intubation
Time Frame: From randomization to Day 28
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CSL312
Number analyzed (Participants) | 61 | 63
percentage of participants | 24.6 | 17.5

4. Secondary Outcome: Number of Participants With ≥ 2-Point Improvement Compared to Baseline on National Institute of Allergy and Infectious Diseases (NIAID) Ordinal Scale
Description: The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 8) Death; 7) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 5) Hospitalized, requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 1) Not hospitalized, no limitations on activities.
Time Frame: From randomization to Day 28
Population: ITT
Measure: Number; unit: participants
Arm/Group | Placebo | CSL312
Number analyzed (Participants) | 61 | 63
participants | 44 | 42

5. Secondary Outcome: Percent of Participants With ≥ 2-Point Improvement Compared to Baseline on NIAID
Description: as for outcome 4
Time Frame: From randomization to Day 28
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CSL312
Number analyzed (Participants) | 61 | 63
percentage of participants | 72.1 | 66.7

6. Secondary Outcome: Number of Participants Within Each of the Categories of the NIAID at End of Study
Description: as for outcome 4
Time Frame: Day 28
Population: ITT
Measure: Number; unit: participants
Arm/Group | Placebo | CSL312
Number analyzed (Participants) | 61 | 63
participants
  Death | 11 | 11
  Hospitalized, on Invasive Mechanical Ventilation or ECMO | 2 | 1
  Hospitalized, on Non-invasive Ventilation or High-flow Oxygen Devices | 2 | 0
  Hospitalized, Requiring Supplemental Oxygen | 1 | 2
  Hospitalized, Not Requiring Supplemental Oxygen - Requiring Ongoing Medical Care | 0 | 0
  Hospitalized, Not Requiring Supplemental Oxygen - no Longer Requiring Medical Care | 0 | 0
  Not Hospitalized, Limitation on Activities and/or Requiring Home Oxygen | 14 | 11
  Not Hospitalized, no Limitations on Activities | 25 | 26
  Not Done | 5 | 6
  Missing | 1 | 6

7. Secondary Outcome: Percent of Participants Within Each of the Categories of the NIAID at End of Study
Description: as for outcome 4
Time Frame: Day 28
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CSL312
Number analyzed (Participants) | 61 | 63
percentage of participants
  Death | 18.0 | 17.5
  Hospitalized, on Invasive Mechanical Ventilation or ECMO | 3.3 | 1.6
  Hospitalized, on Non-invasive Ventilation or High-flow Oxygen Devices | 3.3 | 0
  Hospitalized, Requiring Supplemental Oxygen | 1.6 | 3.2
  Hospitalized, Not Requiring Supplemental Oxygen - Requiring Ongoing Medical Care | 0 | 0
  Hospitalized, Not Requiring Supplemental Oxygen - no Longer Requiring Medical Care | 0 | 0
  Not Hospitalized, Limitation on Activities and/or Requiring Home Oxygen | 23.0 | 17.5
  Not Hospitalized, no Limitations on Activities | 41.0 | 41.3
  Not Done | 8.2 | 9.5
  Missing | 1.6 | 9.5

8. Secondary Outcome: Percent of Participants Requiring Continuous Positive Airway Pressure (CPAP) or Bilevel Positive Airway Pressure (BiPAP)
Time Frame: From randomization to Day 28
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CSL312
Number analyzed (Participants) | 61 | 63
percentage of participants | 16.4 | 19.0

9. Secondary Outcome: Percent of Participants Requiring Extracorporeal Membrane Oxygenation (ECMO)
Description: None of the enrolled subjects required the use of ECMO during their participation in this study. Therefore, no data to report for this outcome measure.
Time Frame: From randomization to Day 28
Population: ITT. None of the enrolled subjects required the use of ECMO during their participation in this study. Therefore, no data to report for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CSL312
Number analyzed (Participants) | 61 | 63
percentage of participants | 0 | 0

10. Secondary Outcome: Percent of Participants Requiring High-Flow Nasal Cannula (HFNC)
Time Frame: From randomization to Day 28
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CSL312
Number analyzed (Participants) | 61 | 63
percentage of participants | 18.0 | 14.3

11. Secondary Outcome: Maximum Change From Baseline in Sequential Organ Failure Assessment (SOFA) Score
Description: The score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems. Each system is scored from 0 (normal function) to 4 (most abnormal) with a total score ranging from 0 to 24. A high total SOFA score have been shown to be related to a worse outcome.
Time Frame: From randomization to Day 28
Population: ITT. Participants with missing values were not included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | CSL312
Number analyzed (Participants) | 50 | 45
score on a scale | 0.5 (1.54) | 0.1 (0.79)

12. Secondary Outcome: Change From Baseline in SOFA Total Score
Description: as for outcome 11
Time Frame: From randomization to Day 28
Population: ITT. Participants with missing values were not included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | CSL312
Number analyzed (Participants) | 15 | 12
score on a scale | -1.0 (1.77) | -1.3 (0.89)

13. Secondary Outcome: Change From Baseline in the Individual Components of SOFA Score
Description: as for outcome 11
Time Frame: From randomization to Day 28
Population: ITT. Participants with missing values were not included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | CSL312
Number analyzed (Participants) | 61 | 63
score on a scale
  Respiration Score: number analyzed (Participants) | 34 | 28
  Respiration Score | -0.6 (1.32) | -1.2 (1.16)
  Coagulation Score: number analyzed (Participants) | 23 | 19
  Coagulation Score | -0.1 (0.42) | 0.4 (1.12)
  Liver Score: number analyzed (Participants) | 21 | 17
  Liver Score | 0.0 (0.22) | 0.0 (0.00)
  Cardiovascular Score: number analyzed (Participants) | 35 | 29
  Cardiovascular Score | 0.4 (1.65) | 0.5 (1.35)
  Central Nervous System Score: number analyzed (Participants) | 26 | 27
  Central Nervous System Score | 0.0 (0.00) | 0.0 (0.19)
  Renal Score: number analyzed (Participants) | 23 | 20
  Renal Score | 0.3 (0.93) | 0.5 (1.10)

14. Secondary Outcome: Length of Hospital Stay
Time Frame: From randomization to Day 28 (+/- 2 days)
Population: ITT
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo | CSL312
Number analyzed (Participants) | 61 | 63
Days | 7.00 [0 to 29] | 6.50 [0 to 28]

15. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Time Frame: Up to 28 days after CSL312 or placebo administration
Population: The Safety Analysis Set (SA) comprises all subjects in the ITT Analysis Set who receive any amount of CSL312 or placebo.
Measure: Number; unit: participants
Arm/Group | Placebo | CSL312
Number analyzed (Participants) | 59 | 58
participants | 40 | 35

16. Secondary Outcome: Percent of Participants Experiencing AEs
Time Frame: Up to 28 days after CSL312 or placebo administration
Population: SA
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CSL312
Number analyzed (Participants) | 59 | 58
percentage of participants | 67.8 | 60.3

17. Secondary Outcome: Number of Participants Experiencing Serious Adverse Events (SAEs)
Time Frame: Up to 28 days after CSL312 or placebo administration
Population: SA
Measure: Number; unit: participants
Arm/Group | Placebo | CSL312
Number analyzed (Participants) | 59 | 58
participants | 19 | 20

18. Secondary Outcome: Percent of Participants Experiencing SAEs
Time Frame: Up to 28 days after CSL312 or placebo administration
Population: SA
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CSL312
Number analyzed (Participants) | 59 | 58
percentage of participants | 32.2 | 34.5

19. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs)
Time Frame: Up to 28 days after CSL312 or placebo administration
Population: SA
Measure: Number; unit: participants
Arm/Group | Placebo | CSL312
Number analyzed (Participants) | 59 | 58
participants | 6 | 5

20. Secondary Outcome: Percent of Participants With AESIs
Time Frame: Up to 28 days after CSL312 or placebo administration
Population: SA
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CSL312
Number analyzed (Participants) | 59 | 58
percentage of participants | 10.2 | 8.6

21. Secondary Outcome: Number of Participants With Anti-CSL312 Antibodies
Time Frame: Up to 28 days after CSL312 or placebo administration
Population: The pharmacodynamic (PD) Analysis Set will comprise all subjects in the Safety Analysis Set who received any amount of CSL312 or placebo and have ≥ 1 blood sample available for analysis of biomarkers.
Measure: Number; unit: participants
Arm/Group | Placebo | CSL312
Number analyzed (Participants) | 59 | 58
participants | 1 | 0

22. Secondary Outcome: Maximum Plasma Concentration (Cmax) of CSL312
Time Frame: Up to 28 days after CSL312 administration
Population: The pharmacokinetic (PK) Analysis Set will comprise all subjects in the Safety Analysis Set who received any amount of CSL312 or placebo and have ≥ 1 blood sample available for CSL312 concentration measurement.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | CSL312
Number analyzed (Participants) | 57
ug/mL | 147.335 (77.1286)

23. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of CSL312
Time Frame: Up to 28 days after CSL312 administration
Population: PK
Measure: Median (Full Range); unit: hours
Arm/Group | CSL312
Number analyzed (Participants) | 57
hours | 0.667 [0.28 to 139.97]

24. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to the Time of the Last Measurable Concentration (AUC0-Last) of CSL312
Time Frame: Up to 28 days after CSL312 administration
Population: PK
Measure: Mean (Standard Deviation); unit: h*ug/mL
Arm/Group | CSL312
Number analyzed (Participants) | 57
h*ug/mL | 15806.644 (9393.6295)

25. Secondary Outcome: Terminal Half-life (T1/2) of CSL312
Time Frame: Up to 28 days after CSL312 administration
Population: PK. Participants with missing values were not included in the analysis.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | CSL312
Number analyzed (Participants) | 9
hours | 226.165 (102.6690)

ADVERSE EVENTS:
Time Frame: Up to 28 days per participant after CSL312 or placebo administration
Description: All-Cause mortality uses ITT set and treatment emergent adverse events uses the safety analysis set.
Arm/Group | Placebo | CSL312
All-Cause Mortality (participants affected / at risk) | 11/61 | 11/63
Serious Adverse Events (participants affected / at risk) | 19/59 | 20/58
Other Adverse Events (participants affected / at risk) | 21/59 | 18/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=59) | CSL312 (N=58)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 6 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 3 (3)
Hypotension (Vascular disorders) | 3 (3) | 1 (1)
Arterial thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 4 (4) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (2)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia escherichia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Brain hypoxia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=59) | CSL312 (N=58)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 5 (5) | 2 (2)
Bradycardia (Cardiac disorders) | 0 (0) | 3 (3)
Transaminases increased (Investigations) | 4 (4) | 1 (1)
Fibrin D dimer increased (Investigations) | 3 (3) | 1 (1)
Hypotension (Vascular disorders) | 6 (6) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 3 (3)
Anxiety (Psychiatric disorders) | 2 (2) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT04409509/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-28): https://cdn.clinicaltrials.gov/large-docs/09/NCT04409509/SAP_001.pdf